CLINICAL TRIAL: NCT03838692
Title: A Study of Ponatinib in Advanced or Metastatic Medullary Thyroid Cancer (MTC)
Brief Title: Ponatinib in Advanced or Metastatic Medullary Thyroid Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed by sponsor
Sponsor: Antonio Fojo (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Antonio Fojo, Assistant Professor of Medicine at the Columbia University Medical, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR5196
Record Dates: First submitted 2019-02-11; First posted 2019-02-12 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Medullary Thyroid Cancer
Keywords: Ponatinib; Metastatic Medullary; Advanced Medullary
MeSH Terms: conditions — Carcinoma, Medullary | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ponatinib Arm (Experimental): Ponatinib tablets will be taken by mouth, continuously, once daily at a dose of 30 mg. A cycle of ponatinib is defined as 28 consecutive days starting with the first day of the treatment cycle. Treatment can be taken with water, with or without food, at approximately the same time each day.
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — A daily oral dose at 30 mg.
  Other Names: ICLUSIG

SUMMARY:
The primary objective of this study is to determine in an exploratory manner the objective overall response rate to ponatinib in the treatment of patients with advanced or metastatic MTC previously treated with cabozantinib or vandetanib who have tumors with rearranged-during-transfection (RET) mutations and have tumors without RET mutations.

DETAILED DESCRIPTION:
Ponatinib is an investigational agent that blocks abnormal cancer proteins and therefore harms cancer cells. It was recently approved by the Food and Drug Administration for leukemia treatment, but is not approved for medullary thyroid cancer treatment. Early studies, however, have shown that medullary thyroid tumors respond to ponatinib. These studies were done in the laboratory and not performed on humans. This is a study designed for patients with medullary thyroid cancer. Treatment will consist of a drug called ponatinib which is a pill that taken once each day and continue throughout the duration of the study. The purpose of the study is to:

1. Determine if this treatment will be effective in decreasing the amount of cancer and, if it does, to determine how long the response will last.
2. Determine the side effects that may occur with this treatment.
3. To analyze genetic mutations in tumors to help us understand how tumors grow and how these drugs interact with the mechanisms within the tumor.

Ponatinib has been given to many patients with leukemia and is now approved by the United States Food and Drug Administration for treatment of certain types of leukemia. This study will seek to determine if ponatinib can bring benefit to patients with medullary thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of localized or metastatic unresectable MTC.
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral computerized tomography (CT) scan.
* The last dose of previous therapy targeting RET kinase must be given at least 4 weeks - Previous treatment with cytotoxic chemotherapy, immunotherapy, or radiotherapy are permitted, if the last dose was given at least 4 weeks prior to the first dose of ponatinib
* Patient must have failed (progressed on or been intolerant of) prior treatment with cabozantinib or vandetanib.
* Age ≥18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Normal organ and marrow function as defined below:
* Negative pregnancy test for women of childbearing potential or male patients, even if surgically sterilized (i.e., status post-vasectomy), who:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or
  * Agree to completely abstain from heterosexual intercourse
* Normal QT interval corrected on screening electrocardiogram (ECG) evaluation, defined as the corrected QT interval by Fredericia (QTcF) of ≤450 ms.
* Ability to understand and the willingness to sign a written informed consent document and follow the guidelines of the clinical protocol including visits for treatment and follow up
* Life expectancy of greater than 12 weeks
* Available archival tissue or willingness to undergo fresh biopsy if no archival tissue is available.

Exclusion Criteria:

* Patients who are receiving any other investigational agent.
* Patients with brain metastases or spinal cord compression unless they completed radiation therapy ≥4 weeks prior to the first dose of ponatinib and are stable without steroids or anti-convulsant therapy for ≥10 days.
* Patients who cannot discontinue medications that are known to be associated with Torsades de Pointes. These medications are listed in Attachment 3
* Uncontrolled hypertension (systolic blood pressure >150 or diastolic blood pressure >100
* Significant or active cardiovascular disease within 6 months prior to enrollment
* A history of pancreatitis or alcohol abuse
* Uncontrolled hypertriglyceridemia (>450 mg/dL)
* Major surgery (with the exception of minor surgical procedures, such as catheter placement or tumor biopsy) within 28 days prior to the first dose of ponatinib
* Ongoing or active infection including known history of human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C (HCV). Testing for these viruses is not required in the absence of a history of infection.
* Suffer from any condition or illness that, in the opinion of the investigator, would compromise patient safety or interfere with the evaluation of the safety of the study drug
* Evidence of a bleeding diathesis that cannot be corrected with standard therapy or factor replacement
* Presence of another primary malignancy within the past 2 years (except for non-melanoma skin cancer or cervical cancer in situ. Prior prostate cancer is also permitted if prostate-specific antigen (PSA) is now undetectable)
* Pregnant or lactating
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  ORR is defined as the proportion of the subjects in the analysis population who have a complete response (CR) or partial response (PR). Responses are based on assessments per RECIST.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 24 months
  PFS is defined as the time from the first day of trial treatment to the first documented disease progression per the Kaplan-Meier curve.

OTHER OUTCOMES:
Total Number of Adverse Reactions | 24 months
  Testing safety and toxicity assessed using CTCAE criteria

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Fojo, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No